CLINICAL TRIAL: NCT07075367
Title: Effect of a Trunk, Hip, Knee and Ankle Exercise Program on Clinical Aspects of People With Diabetic Peripheral Neuropathy: a Randomized Clinical Trial
Brief Title: Effect of an Exercise Program on Clinical Aspects of People With Diabetic Peripheral Neuropathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Piaui (Other)
Responsible Party: Principal Investigator, Vinicius Saura Cardoso, Principal Investigator, Federal University of Piaui
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6.802.243
Record Dates: First submitted 2025-07-11; First posted 2025-07-20 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-07

CONDITIONS: Diabetic Peripheral Neuropathy
Keywords: Diabetic peripheral neuropathy; Exercise therapy; Neuropathy symptoms; Quality of life; Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Blinding will be single-blind, so the outcome evaluator will not be aware of the allocation of participants to the groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proximal/distal protocol (Experimental): The experimental group will receive a proximal/distal exercise program (trunk, hip, knee and ankle).
  Interventions: Other: Proximal/distal protocol
- Distal protocol (Active Comparator): The control group will receive a distal exercise program (ankle and foot) available in the literature and previously tested.
  Interventions: Other: Distal protocol

INTERVENTIONS:
Other: Proximal/distal protocol — The experimental group will receive a proximal/distal exercise program (trunk, hip, knee and ankle) consisting of four stages: warm-up, strengthening, sensorimotor training and relaxation.
  Arms: Proximal/distal protocol
Other: Distal protocol — The control group will receive a distal exercise program available in the literature and previously tested. This will contain warm-up exercises, intrinsic foot muscle strengthening, extrinsic foot-ankle muscle strengthening, and functional exercises.
  Arms: Distal protocol

SUMMARY:
Diabetic Peripheral Neuropathy (DPN) is one of the most prevalent and debilitating complications of type 2 diabetes mellitus (DM2), especially affecting the distal region of the lower limbs. Such changes affect clinical aspects, such as quality of life. Several pieces of evidence point to therapeutic exercises as an effective way to minimize these deficits. This is a single-blind randomized clinical trial in which participants will be randomly assigned to two groups. The stipulated sample size was 64 participants. The experimental group will receive a distal/proximal exercise program and the control group will receive a distal exercise program available in the literature and previously tested. The intervention will last 12 weeks and will take place twice a week, with an average time of 50 minutes. Neuropathic symptoms will be considered primary outcomes. The secondary outcomes evaluated will be: capillary blood glucose, Mini-BESTest, Falls Efficacy Scale (FES), EQ-5D and HADS (depression and anxiety). This study was approved by the local research ethics committee (Opinion 6.802.243), conducted in accordance with the Declaration of Helsinki and in accordance with the CONSORT guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Adult individuals aged between 45 and 75 years, male or female, diagnosed with DM2;
* DPN diagnosis based on vibration sensitivity tests assessed by a 128 Hz tuning fork and tactile sensitivity measured by a 10 g monofilament
* Sedentary or irregularly active individuals (level A) according to the Physical Activity Level Classification - IPAQ
* Score of at least 5 points on the Functional Independence Measure (FIM), i.e., requires supervision, but without physical contact
* Absence of diabetic foot ulcer (DFU) for at least one month
* No amputation or at most amputation of fingers, except for the hallux

Exclusion Criteria:

* Individuals involved in physical training programs simultaneously with the intervention
* History of surgical intervention in the lower limbs or spine
* Use of walking assistance devices
* Diagnosis of severe cardiovascular disorder
* Diagnosis of other neurological impairments in addition to DPN
* Presence of dementia or inability to provide consistent information
* Severe retinopathy

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Symptoms | Baseline (initial assessment, AV1), 12th week (final assessment, AV2) and 16th week (follow up, AV3).
  This consists of 15 "yes/no" questions; 13 items assess symptoms of diabetic peripheral neuropathy, one item assesses peripheral vascular disease (item 4), and one item assesses general asthenia (item 10). "Yes" answers to items 1-3, 5-6, 8-9, 11-12, and 14-15 are each awarded one point. A "no" answer to items 7 and 13 is awarded one point.

SECONDARY OUTCOMES:
Quality of life assessment | Baseline (initial assessment, AV1), 12th week (final assessment, AV2) and 16th week (follow up, AV3).
  The EQ-5D tool will be used, consisting of five questions that assess the following aspects: mobility, personal care, usual activities, pain or discomfort, and anxiety/depression.
Fear of falling | Baseline (initial assessment, AV1), 12th week (final assessment, AV2) and 16th week (follow up, AV3).
  The Falls Efficacy Scale (FES) assesses fear of falling when performing ten easy tasks related to activities of daily living. These 16 activities are scored from one to four. The FES score is the sum of the scores obtained for each item. The total score can range from 16 (no concern) to 64 (extreme concern). Therefore, the lower the score, the greater the confidence, translating into high self-efficacy.
Anxiety and depression level | Baseline (initial assessment, AV1), 12th week (final assessment, AV2) and 16th week (follow up, AV3).
  Hospital Anxiety and Depression Scale. The scale consists of 14 questions that assess how patients felt during the previous week. The questions correspond to a 4-point Likert-type scale, from 0 to 3. Seven of the 14 questions assess the level of depression, and the remaining seven questions assess the level of anxiety, resulting in two subscales with scores ranging from 0 to 21. Higher scores indicate higher levels of anxiety and depression. Additionally, the following categorization can be adopted: 0 to 7 indicating no stress or depression, 8 to 10 indicating moderate levels of anxiety or depression, and >11 indicating high levels of anxiety or depression.
Fall risk | Baseline (initial assessment, AV1), 12th week (final assessment, AV2) and 16th week (follow up, AV3).
  Mini-BESTest. The test includes the domains of anticipatory postural adjustments (up to 6 points), postural responses (up to 6 points), sensory orientation (up to 6 points), and gait stability (up to 10 points). It consists of 14 items scored from 0 to 2, reaching a maximum score of 28, with higher scores corresponding to better postural balance. A private room equipped with the necessary equipment will be used for the test.

IPD SHARING:
Plan to Share IPD: No